CLINICAL TRIAL: NCT02088060
Title: A Four-week, Multicentre, Double-blinded, Randomised, Active- and Placebo- Controlled, Parallel-group Trial Investigating Efficacy and Safety of Cannabidiol in Acute, Early-stage Schizophrenic Patients
Brief Title: A Four-week Clinical Trial Investigating Efficacy and Safety of Cannabidiol As a Treatment for Acutely Ill Schizophrenic Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following the expiry of the original research grant, no follow-up financing could be provided to complete the study.
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other); Heidelberg University (Other); Technical University of Munich (Other); Ludwig-Maximilians - University of Munich (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-FEP; 2012-004335-23 (EudraCT Number)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cannabidiol; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cannabidiol (Experimental): Cannabidiol capsules 2x200 mg twice a day and placebo olanzapine capsule once a day over 4 weeks
  Interventions: Drug: Cannabidiol; Drug: Placebo Olanzapine
- Olanzapine (Active Comparator): Olanzapine capsule 15mg once a day and placebo cannabidiol capsules twice a day over 4 weeks
  Interventions: Drug: Olanzapine; Drug: Placebo Cannabidiol
- Placebo (Placebo Comparator): Placebo cannabidiol capsules twice a day and placebo olanzapine capsule once a day over 4 weeks
  Interventions: Drug: Placebo Cannabidiol; Drug: Placebo Olanzapine

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol capsules
  Arms: Cannabidiol
Drug: Olanzapine — Olanzapine capsules
  Other Names: Olanzapine 1A pharma
  Arms: Olanzapine
Drug: Placebo Cannabidiol — Placebo cannabidiol capsules
  Arms: Olanzapine; Placebo
Drug: Placebo Olanzapine — Placebo olanzapine capsules
  Arms: Cannabidiol; Placebo

SUMMARY:
Schizophrenia is a heterogeneous mental disorder that affects one percent of the world's population. Current antipsychotics are only partially effective, and their use is often associated with serious side effects. Cannabidiol is a natural counterpart of the psychoactive component of marijuana, delta-9-tetrahydrocannabinol. While cannabidiol has no psychotomimetic or addictive properties, it indirectly affects endogenous cannabinoid signalling by impairing the degradation of the endocannabinoid anandamide. In a controlled clinical trial of cannabidiol versus amisulpride (an established antipsychotic) in acute paranoid schizophrenics the investigators showed a significant clinical improvement in all symptoms of schizophrenia compared to baseline with either treatment. But cannabidiol displayed a significantly superior side-effect profile. This study is to evaluate the efficacy and safety of this novel treatment option in comparison to placebo and olanzapine, an established second generation antipsychotic in the treatment of acute schizophrenia and schizophrenia maintenance therapy, in a four-week clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the subject
* DSM-IV-TR diagnosis of schizophrenic psychosis (295.10, 295.20, 295.30, 295.90 (American Psychiatric Association)
* Patients must be within the first three years of illness, i.e. first diagnosis of schizophrenia is no older than three years.
* Age 18 to 65 years, male or female
* Minimal initial PANSS score of 75 at baseline
* Female patients of childbearing potential need to utilize a proper method of contraception.
* Body Mass Index between 18 and 40

Exclusion Criteria:

* Lack of accountability (assessed by an independent psychiatrist)
* History of treatment-resistant schizophrenia, defined as no response to at least two antipsychotics given for a minimum of 6 weeks each in an adequate dosage
* Positive urine drug-screening for illicit drugs at screening (except cannabinoids and benzodiazepines)
* Serious suicidal risk at screening visit (Subject to investigator's and independent psychiatrist's judgement: Poses a serious suicidal or homicidal risk at screening visit or has made a serious suicide attempt within the last 12 months prior to screening visit, or has exhibited homicidal behaviour at anytime during her/his lifetime)
* Known intolerance or allergy to olanzapine or cannabidiol
* Other relevant interferences of axis 1 (e.g. serious depression) according to diagnostic evaluation (MINI) including residual forms of schizophrenia
* Pregnancy, as determined through a β-HCG pregnancy test, or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-12-08 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Change in the Positive and Negative Syndrome Scale (PANSS) total score | within 4 weeks

SECONDARY OUTCOMES:
Changes in the PANSS subscores and clusters | within 4 weeks
Changes in the Clinical Global Impression score | within 4 weeks
Changes in the Global Assessment of Functioning Scale | within 4 weeks
Changes in the Personal and Social Performance Scale | within 4 weeks
Changes in the Calgary Depression Scale for Schizophrenia | within 4 weeks
Changes in the Hamilton Anxiety Scale | within 4 weeks
Changes in cognitive skills | within 4 weeks
Response to antipsychotic medication | within 4 weeks
Plasma levels of endogenous cannabinoids | within 4 weeks
Changes in physiological parameter | within 4 weeks
Changes in the UKU Side Effect Rating Scale | within 4 weeks
Columbia Suicidality Severity Rating Scale | within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: F. Markus Leweke, MD, Principal Investigator — Central Institute of Mental Health
Locations (6):
- Psychiatric Centre Glostrup, Glostrup Municipality, Denmark
- Germany (5):
  - Department of General Psychiatry, Heidelberg University, Heidelberg, Baden-Wurttemberg
  - Dep. of Psychiatry and Psychotherapy, Central Institute of Mental Health, Mannheim, Baden-Wurttemberg
  - Dept. of Psychiatry and Psychotherapy, Ludwig-Maximillians-University Munich, Munich, Bavaria
  - Dept. of Psychiatry and Psychotherapy, Technical University Munich, Munich, Bavaria
  - Dept. of Psychiatry and Psychotherapy, Martin-Luther-University, Halle/Wittenberg, Halle, Saxony-Anhalt